CLINICAL TRIAL: NCT03686059
Title: Outcome of Concomitant Use of Punctal Plugs and Omeg 3 Fatty Acids on Ocular Surface Disease in Patients Using Systemic Isotretinoin
Brief Title: Outcome of Omega 3 FA and Punctal Plugs on Ocular Surface Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer of ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hamaky1
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Ocular Surface Disease
MeSH Terms: interventions — Docosahexaenoic Acids; Punctal Plugs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- punctal plug (Experimental): SOFT PLUG® Preloaded Silicone Plugs by OASIS®
  Interventions: Device: punctal plug
- Combined (Experimental): SOFT PLUG® Preloaded Silicone Plugs by OASIS® plus Daily intake of DHA (docosahexaenoic acid)
  Interventions: Drug: Omega 3; Device: punctal plug
- control (No Intervention): no medication was given

INTERVENTIONS:
Drug: Omega 3 — daily intake of 250 mg
  Other Names: docosahexaenoic acid
  Arms: Combined
Device: punctal plug — punctal plug will be inserted in inferior punctum
  Other Names: OASIS SOFT PLUG
  Arms: Combined; punctal plug

SUMMARY:
Ocular surface disease is a common adverse effect of systemic isotretinoin therapy.

The investigators consider that punctal plugs and Omega 3 is a good line for treatment of ocular surface disease associated with systemic isotretinoin therapy

DETAILED DESCRIPTION:
Subjective and objective evaluation of ocular surface disease was done at baseline ,1 and 3 months of the study .

ELIGIBILITY:
Inclusion Criteria:

* systemic isotretinoin therapy

Exclusion Criteria:

* systemic or ocular diseases ,previous ocular surgery, corneal pathology and contact lens wearer

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Break up Time at baseline and during the study | 3 months
  fluorescein sodium stripes will be used for measurement of Break up Time in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- ACDS, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided